CLINICAL TRIAL: NCT04204759
Title: The Effect of Transcranial Direct Current Stimulation of the Prefrontal Cortex on Antisocial Behavior
Brief Title: Transcranial Direct Current Stimulation and Antisocial Behavior
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nanyang Technological University (Other)
Responsible Party: Principal Investigator, Olivia Choy, Assistant Professor, Nanyang Technological University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB-2019-06-072
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Aggression
Keywords: transcranial direct curren stimulation; antisocial behavior
MeSH Terms: conditions — Aggression; Antisocial Personality Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anodal stimulation (Experimental): Participants in the active stimulation group will undergo anodal transcranial direct current stimulation (tDCS). tDCS will be delivered by a battery-driven, constant-current stimulator connected to two saline-soaked surface sponge electrodes. An anodal electrode (25cm2) will be placed over the ventromedial prefrontal cortex and one cathodal electrode (35cm2) will be placed over the occipital cortex. Scalp electrodes will be positioned according to the 10-20 EEG international system. A current of 2mA will be applied for 20 minutes and the current will be ramped up and down over 30 seconds at the beginning and end of the stimulation period.
  Interventions: Device: Transcranial direct current stimulation
- Sham stimulation (Sham Comparator): The sham tDCS condition will involve the same placement of the electrodes, current intensity, and ramp-up/down time as the active tDCS condition, but stimulation will only last for 30 seconds.
  Interventions: Device: Sham transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Non-invasive stimulation will be conducted using a tDCS device (StarStim, Neuroelectrics, Spain).
  Arms: Anodal stimulation
Device: Sham transcranial direct current stimulation — The same device will be used as in the active stimulation group, but stimulation will be terminated after 30 seconds.
  Arms: Sham stimulation

SUMMARY:
The main objective of this study is to investigate the causal relationship between prefrontal cortex activity and antisocial behavior, as well as risk factors for antisocial behavior. Specifically, this study tests the hypothesis that upregulating activity in the prefrontal cortex through a non-invasive form of brain stimulation, transcranial direct current stimulation (tDCS) will reduce antisocial and aggressive behavior. The effects of 3 days of anodal stimulation over the prefrontal cortex are assessed.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 (with parental consent) or above 21 (without parental consent)
* Able to understand the nature of the study and give informed consent

Exclusion Criteria:

* History of or active neurologic, cardiovascular, or psychiatric disease including anxiety disorders (e.g., PTSD, panic attacks, obsessive-compulsive disorder) and mood disorders (e.g., depression)
* Currently consuming anti-convulsant, anti-psychotic, or sedative/hypnotic medications
* Currently consuming anti-depressants
* History of seizures
* Metallic implants on scalp
* Participated in any other non-invasive brain stimulation study in the same day
* Ever had an adverse reaction to tDCS

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2019-11-03 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Points in the Point Subtraction Aggression Paradigm after stimulation | Within 1 hour after the third consecutive active tDCS or sham session
  The number of points earned on the lab task will be assessed.
Antisocial behavior inclinations after stimulation | Within 1 hour after the third consecutive active tDCS or sham session
  This will be assessed using 5 hypothetical scenarios in which someone commits a criminal or antisocial act. Participants will respond to the likelihood that they would commit the act in the scenario according to a 10-point Likert scale. Responses are measured on a scale ranging from zero (no chance at all) to 10 (100% chance). A higher value reflects a greater intention to engage in the antisocial act.
Moral judgment ratings after stimulation | Within 1 hour after the third consecutive active tDCS or sham session
  This will be assessed using 5 hypothetical scenarios in which someone commits a criminal or antisocial act. Participants will rate the moral wrongfulness of the act in the scenario on a scale from 0 (not at all) to 10 (very). A higher score reflects a greater perception of moral wrongfulness regarding the antisocial act.
Delay discounting rates after stimulation | Within 1 hour after the third consecutive active tDCS or sham session
  Participants' responses to 5 questions indicating if they would prefer a smaller reward today or a larger reward in the specified number of days will be assessed. The delay discount rates (k) of monetary rewards will be calculated based on the responses to the 5 trials.
Helping behavior after stimulation | Within 1 hour after the third consecutive active tDCS or sham session
  This will be assessed based on the number of easy and hard puzzles participants choose to assign to another participant in the study.
Antisocial behavior after stimulation | Within 1 hour after the third consecutive active tDCS or sham session
  This will be assessed based on the participants' accurate reporting of the number of problems correctly solved in a task.

SECONDARY OUTCOMES:
Number of participants with adverse events | Within 1 hour after each of the 20-minute active tDCS or sham sessions
  The number of participants reporting the experience of sensations resulting from tDCS will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Olivia Choy, PhD, Principal Investigator — Nanyang Technological University
Locations (1):
- Nanyang Technological University, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No